CLINICAL TRIAL: NCT04155515
Title: A Phase III, Multicenter, Open-labeded Study To Evaluate Efficacy and Safety of TG-2349 in Combination With DAG181 and Ribavirin for 12 Weeks of Treatment in HCV Genotype I Infected Patients
Brief Title: A Phase III Study to Evaluate Efficacy and Safety of TG-2349 in Combination With DAG181 and RBV for HCV Type I Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dongguan HEC TaiGen Biopharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TGDAG-C-3
Record Dates: First submitted 2019-11-05; First posted 2019-11-07 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-01

CONDITIONS: Chronic Hepatics C Virus (HCV) Genotype 1; Non-Cirrhotic; Cirrhosis; Treatment naïve
Keywords: Chronic Hepatics C Virus (HCV) Genotype 1; Non-Cirrhotic; Cirrhosis; Treatment naïve; efficacy; safety; TG-2349; DAG181; Ribavirin
MeSH Terms: conditions — Hepatitis C; Fibrosis | interventions — yimitasvir; Ribavirin

STUDY DESIGN:
Intervention Model Description: The non-cirrhotic, HCV genotype 1 infected subjects will be assigned to Group 1. The cirrhotic, HCV genotype 1 infected subjects will be assigned to Group 2. The subjects in Group 1 and 2 will be treated with TG-2349 400mg combined with DAG181 200mg and Ribaverin 1000mg/1200mg for 12 weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-cirrhotic, HCV genotype 1 infected subjects (Other): Subjects will be treated with TG-2349 400mg combined with DAG181 200mg and Ribaverin 1000mg/1200mg for 12 weeks.
  Interventions: Drug: TG-2349; Drug: DAG181; Drug: Ribavirin
- Cirrhotic, HCV genotype 1 infected subjects (Other): Subjects will be treated with TG-2349 400mg combined with DAG181 200mg and Ribaverin 1000mg/1200mg for 12 weeks.
  Interventions: Drug: TG-2349; Drug: DAG181; Drug: Ribavirin

INTERVENTIONS:
Drug: TG-2349 — TG-2349 400mg
Drug: DAG181 — DAG181 200mg
Drug: Ribavirin — Ribavirin 1000mg/1200mg

SUMMARY:
A Phase III, Multicenter, open-labeded study to Evaluate Efficacy and Safety of TG-2349 in Combination With DAG181 and Ribavirin for 12 weeks of treatment in HCV Genotype I Infected Patients

DETAILED DESCRIPTION:
The purpose of this study is to evaluate efficacy and safety of TG-2349 in combination with DAG181 and Ribavirin for 12 weeks of treatment in HCV Genotype I infected patients. Approximately 360 subjects will be enrolled in this study and divided into 2 groups:

Group 1: Chronic hepatics C virus (HCV) genotype 1 infected, non-cirrhotic subjects.

Group 2: Chronic hepatics C virus (HCV) genotype 1 infected, cirrhotic subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Before starting the study, an informed consent form (ICF) approved by the Institutional Review Board (IRB) is obtained from the subject or his/her legal representative；
2. Male or female, and ≥18 years of age inclusive when signing ICF；
3. Body mass index (BMI) in the range of 18.0 to 35.0kg/m2 and body weight ≥ 40 kg at Screening；
4. Presence of chronic hepatitis C (CHC) as documented below: (1)A positive anti-HCV antibody test or positive HCV RNA or positive HCV genotyping test at least 6 months prior to the Baseline/Day 1 visit or, (2) A liver biopsy performed prior to the Baseline/Day 1 visit with evidence of chronic HCV infection；
5. Positive for anti-HCV antibody at Screening；
6. Presence of an HCV RNA level ≥ 1 x 10^4 IU/mL at Screening as determined by the Central Laboratory；
7. Presence of genotype 1a, 1b, or 1a/1b combination HCV-infection at Screening as determined by the Central Laboratory；
8. HCV treatment naïve defined as no prior therapy with any interferon (IFN), ribavirin (RBV), or other approved or investigational HCV-specific agent；
9. Without or with cirrhosis: (1) Without cirrhosis as defined as any one of the following: (a) Liver biopsy without showing cirrhosis (e.g., Metavir score < F4 or Ishak score < 5) within one year prior to Screening or at Screening. (b) FibroScan showing cirrhosis or results ≤ 12.5 kPa within six months prior to Screening or at Screening. (2) With cirrhosis as defined as any one of the following: (a) Liver biopsy showing cirrhosis (e.g., Metavir score = F4 or Ishak score ≥ 5) within one year prior to Screening or at Screening. (b) FibroScan showing cirrhosis or results > 12.5 kPa within six months prior to Screening or at Screening；NOTICE: If there is liver biopsy, liver biopsy results will supersede non-invasive testing results and be considered definitive.
10. ECG without clinically significant abnormalities at Screening；
11. Subjects must have the following laboratory parameters at Screening: (1) ALT ≤ 10 × the upper limit of normal (ULN). (2) AST ≤ 10 × ULN. (3) Without cirrhosis: Total bilirubin ≤ 1.5 × ULN except history of Gilbert's syndrome. If Gilbert's syndrome is the proposed etiology, the total bilirubin must ≤ 2 × ULN. With cirrhosis: Total bilirubin ≤ 2 × ULN. (4) Platelet count ≥ 90,000 cells/mm3. (5) Absolute neutrophil count (ANC) ≥ 1,500 cells/mm3. (6) HbA1c ≤ 8.5%. (7) Creatinine clearance (CLcr) ≥ 50 mL /min, as calculated by the Cockcroft-Gault equation. (8) Hemoglobin ≥ 110 g/L for female subjects; ≥ 120 g/L for male subjects. (9) Without cirrhosis Albumin ≥ 3.5 g/dL；With cirrhosis Albumin ≥30g/L. (10) Without cirrhosis INR ≤ 1.5 x ULN；With cirrhosis INR ≤ 1.7 x ULN. (11) Alpha fetoprotein (AFP)<100 ng/mL；20ng/mL≤AFP≤100ng/mL need to take Liver Ultrasonic testing to exclude subjects with suspicious liver cancer cells. (12) Anti-nuclear antibodies (ANA) ≤ 1:320；
12. A female subject is eligible to enter the study if it is confirmed that she is: (1) Of non-childbearing potential (i.e., women who have had a hysterectomy, have both ovaries removed or medically documented ovarian failure, or are postmenopausal - women > 50 years of age with cessation (for ≥12 months) of previously occurring menses), or (2) Of childbearing potential (Women ≤ 50 years of age with amenorrhea will be considered to be of childbearing potential). These women must have a negative serum pregnancy test at Screening and agree to consistently and correctly use an approved contraceptive method (i.e. abstinence, vaginal ring, cervical cap, contraceptive diaphragm, or intrauterine devices) from screening until at least 6 months after the last dose of study drug(s)；
13. Male subjects must agree to consistently and correctly use an approved contraceptive method (i.e. abstinence, condom, or spouses using contraceptive drugs, vaginal ring, cervical cap, contraceptive diaphragm, or intrauterine devices) from screening until at least 6 months after the last dose of study drug(s)；
14. Male subjects must agree to refrain from sperm donation from screening until at least 6 months after the last dose of study drug(s)；
15. Subject must be of generally good health, with the exception of chronic HCV infection, as determined by Investigator；
16. Subject must be able to comply with the dosing instructions for study drug administration and able to complete the study schedule of assessments, including all required post-treatment visits.

Exclusion Criteria:

1. Positive serological test for IgM anti-HAV or anti-HEV antibody at Screening；
2. Positive serological test for HBsAg at Screening；
3. Positive test for HIV-1 or HIV-2 at Screening；
4. Clinically-relevant drug abuse within 12 months of signing the ICF. A positive drug screen will exclude subjects unless it can be explained by a prescribed medication; the diagnosis and prescription must be approved by Investigator；
5. Alcohol misuse as defined by an AUDIT score of ≥ 8；
6. Contraindications to RBV therapy, including hemoglobinopathies (e.g., thalassemia major or sickle-cell anemia)；
7. Pregnant or nursing female or male with pregnant female partner；
8. Use of any prohibited medications before Baseline/Day 1 visit；
9. Known hypersensitivity to TG-2349, DAG181, RBV, sulfa drugs, or formulation excipients；
10. Current or prior history of any of the following: (1) Chronic hepatic disorder not induced by HCV (including but not limited to Hemochromatosis, Wilson's disease, alpha-1 antitrypsin deficiency, cholangitis, autoimmune hepatitis, alcoholic liver disease, drug-induced liver disease. (2) Decompensated liver cirrhosis (Child-Pugh class B and C). (3) Any dysphagia, malabsorption syndrome, or other gastrointestinal disturbances affecting drug absorption. (4) Difficulty with blood collection and/or poor venous access for the purposes of phlebotomy. (5) Central nervous system (CNS) trauma, seizure disorder, stroke or transient ischemic attack. (6) Solid organ transplantation. (7) Significant cardiac disease (including but not limited to the myocardial infarction based on ECG and/or clinical history). (8) Significant pulmonary disease or porphyria (e.g. lung infiltration or impaired lung function). (9) Pancreatitis. (10) Autoimmune disease (systemic lupus erythematosus, rheumatoid arthritis, sarcoidosis, psoriasis). (11) Psychiatric hospitalization, suicide attempt, and/or a period of disability as a result of their psychiatric illness within the last 5 years. (12) Malignancy within 5 years prior to Screening, with the exception of specific cancers that are entirely cured by surgical resection (basal cell skin cancer, etc). Subjects under evaluation for possible malignancy are not eligible. (13) Serious acute drug allergy (such as anaphylaxis or hepatotoxicity) or serious skin hypersensitive reaction (such as vesicular rash, Stevens Johnson Syndrome)；
11. As determined by Investigator, a subject that would affect the therapy, evaluation or compliance with the protocol is not suitable to take part in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 370 (Actual)
Dates: Start 2019-06-13 (Actual); Primary Completion 2020-08-11 (Actual); Study Completion 2020-08-11 (Actual)

PRIMARY OUTCOMES:
The proportion of antiviral efficacy (HCV RNA < lower limit of quantification, target detected or target not detected) at 12 weeks after the end of treatment | 12 weeks after the end of treatment
  To evaluate the antiviral efficacy

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tsinghua Changgung Hospital, Beijing, China